CLINICAL TRIAL: NCT03758209
Title: Comparison of Preoperative Multimodal Preparation Program (Prehabilitation) With Enhanced Recovery Program for Elective Colorectal Cancer Surgery.
Brief Title: Prehabilitation Versus Enhanced Recovery Program for Elective Colorectal Cancer Surgery.
Acronym: PrehabVsERAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Borbala Hospital (Other Government)
Collaborators: St. Borbala Hospital, Department of Surgery (Unknown); Semmelweis University (Other)
Responsible Party: Principal Investigator, Dr. Balázs Bánky PhD, Head of the Department of Surgery, St. Borbala Hospital, St. Borbala Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 48931-2/2018/EKU ETT-TUKEB
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Colorectal Cancer; Insulin Resistance
Keywords: Morbidity, Mortality, Complication, Prehabilitation, ERAS
MeSH Terms: conditions — Colorectal Neoplasms; Insulin Resistance | interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: Patients planned for elective, curative operations for colorectal cancer will be randomized into two groups: experimental group will take part in a dedicated 4-week multimodal preparation program followed by ERAS preoperative management, while control group will just participate in the ERAS program without specific physical and mental preparation.
  1:1 randomization will be performed.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators and assessors will be blinded regarding preoperative preparation. Both randomization process and rehabilitation process will be carried out by a trained nurse, physiotherapist and psychotherapist, neither of them will be involved in outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation + ERAS (Experimental): Patients receiving a formal preoperative preparation on:
  * Physical status (walking, respiratory training)
  * Nutrition (nutritional supplements)
  * Mental status (weekly groups led by clinical psychologist on anxiety and depression management).
  Each patient will be treated in an ERAS program preoperatively.
  Interventions: Procedure: Prehabilitation + ERAS; Procedure: ERAS
- ERAS (Active Comparator): Each patient will be treated in an ERAS program preoperatively. No specific preoperative training will be involved apart from nutritional status assessment and nutritional supplements.
  Interventions: Procedure: ERAS

INTERVENTIONS:
Procedure: Prehabilitation + ERAS — Prehabilitation will cover a range preoperative education and exercises (weekly) on diet, physical activity (daily walking), respiratory training (forced deep inspiration with spirometer device), as well as anxiolytic group psychotherapy.
  Arms: Prehabilitation + ERAS
Procedure: ERAS — Enhanced Recovery Program, including preoperative 4 weeks nutritional supplementation.
  Other Names: Enhanced Recovery After Surgery Program

SUMMARY:
Elective surgery is the most effective treatment option for colorectal cancer, however it has been recognized to be associated with high morbidity and mortality risks.

ERAS (Enhanced Recovery After Surgery) is a preoperative multimodality treatment package, which has been well investigated and proved to be effective in reducing early postoperative morbidity, mortality, length of hospital stay and hospital costs, as well. Still, a good proportion of patients are not suitable for ERAS program, mainly based on lack of compliance and the impaired physical function before surgery.

Prehabilitation Program is a recently introduced trimodal preoperative preparation (training) program, which addresses improvement of physical, mental and nutritional status of the high risk elective surgery patients.

This study aims to investigate the benefit of all efforts of a 4-6-week preoperative preparation program (Prehabilitation) being added to an established ERAS protocol.

DETAILED DESCRIPTION:
Aim:

Colorectal cancer patients with a planned resection are tested if a complex, trimodal rehabilitation program can hold functional and morbidity benefit for them.

In the prospective, randomized (1:1) study control patient group will be the well established and tested ERAS (enhanced recovery after surgery) Program.

Study protocol in details:

1. First visit: Outpatient Department of Surgery

   On both arms:

   • History taking (including family history and oncologic history);

   • Physical examination
   * Operation indication, type of procedure and date of procedure agreed;
   * Organizing further investigations, anesthesia;
   * Operative risk assessment ("ACS - surgical risk calculator");
   * Study patient identifier Nr generated;
2. Nurse-led ERAS/Prehab clinic: randomization

   On both arms:

   • Randomization (Prehabilitation Program / ERAS Program).

   • Nurse led clinic assessment ("study nurse"): .i. CaseReportForm (CRF) filled in.

   .ii. Patient data (personal data, demographics, history) .iii. Anthropometrics (BMI, MUST, Body fat % measurement). .iv. Mental hygienic status assessment (smoking, alcohol consumption, anxiety, depression, sleeping disorders).

   .v. Cardiovascular status (resting HR, RR). .vi. Operative risk assessment (CR-Possum score). .vii. Preoperative counseling (operation type, preparation, pain management, discharge plan).

   .viii. Preoperative nutritional planning (education, nutrient prescription). .ix. Alcohol intake and smoking cessation - information given. .x. Stoma education started. .xi. Consent signed, patient workbook handed over. .xii. Respiratory test referral.
3. Physiotherapy, first visit

   Both on control and interventional arms:
   * Respiratory function test recorded.
   * Physical status tested (6MWD) on a treadmill.

   Just on Prehabilitation arm:

   • Respiratory training education.

   • Respiratory trainer device usage educated.

   • Daily activity (walking) planned.
4. Physiotherapy - second/third/fourth visit (weekly)

   Just on Prehabilitation arm:
   * Previous week activity reviewed as to workbook.
   * Physical assessment: 6MWD, FVC.
   * Next week activity planned.
5. Psychic preparation

   Just on Prehabilitation arm:

   • Once a week half an hour group relaxation training - regardless of the stage of prehabilitation program.
6. Admission to the Surgical Ward a day before surgery

   Both on control and interventional arm:

   • Preoperative assessment: .i. Anthropometrics (BMI, body fat%). .ii. Cardiovascular stage (resting HR and RR), ECG. .iii. Respiratory function tests.

   .iv. Physical status (6MWD) .v. Mental status (Hospital Anxiety and Depression Scale (HADS)) assessment.

   • Preoperative preparation (as to ERAS protocol).

   • Postoperative care (ITU, pain management, mobilization, oral nutrition built up, drains early removal, complications recorded (Clavien-Dindo-classification)).

   • Stoma education.
   * Dietary education.
   * On discharge: Quality of Life (QoL) SF36 - (36-Item Short Form Survey from the RAND Medical Outcomes Study).
7. Postoperative follow up:

Both on control and interventional arms:

• Assessment (4th and 8th week post op.):

.i. Anthropometrics (BMI, Body fat %) .ii. Cardiovascular status (resting HR and RR). .iii. Respiratory function tests. .iv. Physical status (6MWD).

ELIGIBILITY:
Inclusion Criteria:

* patient with histologically proven primary colorectal adenocarcinoma
* any stage of colorectal cancer
* elective operation
* curative intention
* informed consent signed by patient

Exclusion Criteria:

* emergency operation
* palliative operation
* non-colorectal, second malignancy
* pregnancy
* patient not giving consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | within 45 days
  Postoperative length of hospital stay in days.
Number of days spent on ICU (Intensive care unit). | within 45 days postoperative
  Number of days observed on ICU right after operation.
Morbidity (early) classified after Clavien-Dindo. | 7 days (until 8th postoperative day) postoperative
  7-day morbidity will be detailed assessed. Grade 3 or above morbidity rate will be assessed.
Morbidity (long term) classified after Clavien-Dindo. | 30 days (until 31st postoperative day)
  30-day morbidity will be detailed assessed. Grade 3 or above morbidity rate will be assessed.
30-day mortality | 30 days postoperative
  30-day mortality of each patient will be recorded.
90-day mortality | 90 days postoperative
  90-day mortality of each patient will be recorded.
Change in preoperative functional status - 6MWD by operation | Measured points: 4 weeks before surgery, on day of hospital admission
  6MWD (6-minute walking distance test)
Change in postoperative functional status - 6MWD by the end of rehabilitation | Measured points: 4 weeks before surgery, 8 weeks after operation
  6MWD (6-minute walking distance test)
Change in preoperative functional status - FVC by operation | Measured points: 4 weeks before surgery, on day of hospital admission
  FVC (forced vital capacity) will be measured.
Change in preoperative functional status - FVC by the end of rehabilitation | Measured points: 4 weeks before surgery, 8 weeks after operation
  FVC (forced vital capacity) will be measured.

SECONDARY OUTCOMES:
Delay in beginning of adjuvant oncotherapy (chemotherapy, radiotherapy). | within 8 weeks, if adjuvant oncotherapy is needed
  Sufficient recovery time until fitness of adjuvant chemo/radiotherapy will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Balázs Bánky, PhD, Study Director — Department of Surgery, St. Borbala Hospital
Locations (1):
- Department of Surgery, St. Borbala Hospital, Tatabánya, Hungary

REFERENCES:
- [Background] Souwer ETD, Bastiaannet E, de Bruijn S, Breugom AJ, van den Bos F, Portielje JEA, Dekker JWT. Comprehensive multidisciplinary care program for elderly colorectal cancer patients: "From prehabilitation to independence". Eur J Surg Oncol. 2018 Dec;44(12):1894-1900. doi: 10.1016/j.ejso.2018.08.028. Epub 2018 Sep 8. PMID 30266205
- [Background] Bousquet-Dion G, Awasthi R, Loiselle SE, Minnella EM, Agnihotram RV, Bergdahl A, Carli F, Scheede-Bergdahl C. Evaluation of supervised multimodal prehabilitation programme in cancer patients undergoing colorectal resection: a randomized control trial. Acta Oncol. 2018 Jun;57(6):849-859. doi: 10.1080/0284186X.2017.1423180. Epub 2018 Jan 12. PMID 29327644
- [Background] Chen BP, Awasthi R, Sweet SN, Minnella EM, Bergdahl A, Santa Mina D, Carli F, Scheede-Bergdahl C. Four-week prehabilitation program is sufficient to modify exercise behaviors and improve preoperative functional walking capacity in patients with colorectal cancer. Support Care Cancer. 2017 Jan;25(1):33-40. doi: 10.1007/s00520-016-3379-8. Epub 2016 Aug 18. PMID 27539131
- [Background] Carli F, Silver JK, Feldman LS, McKee A, Gilman S, Gillis C, Scheede-Bergdahl C, Gamsa A, Stout N, Hirsch B. Surgical Prehabilitation in Patients with Cancer: State-of-the-Science and Recommendations for Future Research from a Panel of Subject Matter Experts. Phys Med Rehabil Clin N Am. 2017 Feb;28(1):49-64. doi: 10.1016/j.pmr.2016.09.002. PMID 27913000
- [Background] Banky B, Lakatos M, Varga K, Hansagi E, Horvath E, Jaray G. [Enhanced Recovery Program in colorectal surgery]. Magy Seb. 2018 Mar;71(1):3-11. doi: 10.1556/1046.71.2018.1.1. Hungarian. PMID 29536753